CLINICAL TRIAL: NCT00559585
Title: A Phase IIIB Multicenter, Randomized, Double-Blind, Double-Dummy Study to Compare the Efficacy and Safety of Abatacept Administered Subcutaneously and Intravenously in Subjects With Rheumatoid Arthritis, Receiving Background Methotrexate, and Experiencing an Inadequate Response to Methotrexate
Brief Title: Methotrexate-Inadequate Response Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-174; EUDRACT # 2007-005434-37
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Injections, Subcutaneous; Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous (SC) Abatacept (Active Comparator): Participants received 125 mg weekly SC abatacept injections (with an intravenous [IV] abatacept loading dose on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV Placebo) with the exception that on Day 1 a loading dose of IV abatacept replaced the IV Placebo treatment.
  Interventions: Drug: Subcutaneous (SC) Abatacept
- Intravenous (IV) Abatacept (Active Comparator): Participants received IV abatacept infusions on Days 1, 15, 29, and every 28 days, thereafter. A double-dummy design was used to protect the blind, thus, participants also received SC injections of placebo (SC Placebo).
  Interventions: Drug: Intravenous (IV) Abatacept

INTERVENTIONS:
Drug: Subcutaneous (SC) Abatacept — Participants received 125 mg weekly SC abatacept injections (with an intravenous [IV] abatacept loading dose on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV Placebo) with the exception that on Day 1 a loading dose of IV abatacept replaced the IV Placebo treatment.
  Other Names: Orencia; BMS-188667
  Arms: Subcutaneous (SC) Abatacept
Drug: Intravenous (IV) Abatacept — Participants received IV abatacept infusions on Days 1, 15, 29, and every 28 days, thereafter. A double-dummy design was used to protect the blind, thus, participants also received SC injections of placebo (SC Placebo).
  500mg (for body weight up to 60 kg)
  750 mg (body weight between 61 and 100 kg)
  1g (body weight above 100 kg)infusions
  Other Names: Orencia; BMS-188667
  Arms: Intravenous (IV) Abatacept

SUMMARY:
The purpose of this study is to determine whether a weekly subcutaneous dose of abatacept yields clinical efficacy comparable to that of monthly intravenous doses of abatacept in participants with rheumatoid arthritis and an inadequate response to current methotrexate therapy.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects who are considered methotrexate inadequate responders
* 10 or more swollen joints (66 joint count) and 12 or more tender joints (68 joint count)

Exclusion Criteria:

* Subjects who failed one or multiple anti-tumor necrosis factor (TNF) therapies
* Subjects who meet diagnostic criteria for any other rheumatic disease (e.g., lupus erythematous)
* Subjects with active vasculitis of a major organ system (except for subcutaneous rheumatoid nodules)
* Subjects with severe chronic or recurrent bacterial infections
* Subjects who have received treatment with rituximab

An Anti-TNF Failure Sub-study was initiated (recruited separately from Main study) using the same treatment as the Main study in order to assess the immunogenicity and safety in the Anti-TNF Failure population. The Sub-study terminated due to low recruitment and participants were permitted to roll into the LT Open Label Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2492 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (175):
- United States (70):
  - Rheumatology Associates, Pc, Birmingham, Alabama
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Advanced Arthritis Care & Research, Scottsdale, Arizona
  - Catalina Pointe Clinical Research, Inc., Tucson, Arizona
  - St. Joseph'S Mercy Clinic, Hot Springs, Arkansas
  - Talbert Medical Group, Huntington Beach, California
  - Allergy & Rheumatology Medical Clinic, Inc., La Jolla, California
  - Valerius Medical Group &Research Ctr. Of Greater Long Beach, Long Beach, California
  - Stanford University School Of Medicine, Palo Alto, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Boulder Medical Center, Boulder, Colorado
  - Arthritis Assoc And Osteo Ctr Of Col Sprgs, Colorado Springs, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - Arthritis Center Of The Rockies, Pc, Loveland, Colorado
  - Guadagnoli, Germano, Bridgeport, Connecticut
  - Joao Nascimento, Bridgeport, Connecticut
  - Clinical Research Center Of Ct/Ny, Danbury, Connecticut
  - Arthritis And Rheumatic Disease Specialties, Aventura, Florida
  - Arthritis & Osteoporosis Treatment Center, Pa, Orange Park, Florida
  - Rheumatology Associates Of Central Florida, Orlando, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Arthritis & Rheumatology Of Georgia,Pc, Atlanta, Georgia
  - Boise Rheumatology/ Intermountain Research Center, Inc, Boise, Idaho
  - Coeur D'Alene Arthrit Clin, Coeur d'Alene, Idaho
  - Quincy Medical Group, Quincy, Illinois
  - Rockford Orthopedic Associates, Ltd., Rockford, Illinois
  - The Arthritis Center, Springfield, Illinois
  - Klein And Associates, M.D., Pa, Cumberland, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Shores Rheumatology, P. C., Saint Clair Shores, Michigan
  - Arthritis Assoicates Of Mississippi, Jackson, Mississippi
  - Kansas City Internal Medicine, Lee's Summit, Missouri
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Allergy And Arthritis Associates, Dover, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Albuquerque Rehabilitation & Rheumatology Pc, Albuquerque, New Mexico
  - The Center For Rheumatology, Llp, Albany, New York
  - Southern Tier Arthritis & Rheumatism, Olean, New York
  - Arthritis Health Associates, Syracuse, New York
  - Asheville Rheumatology & Osteoporosis Research Asso P. A., Asheville, North Carolina
  - The Arthritis Clinic & Carolina Bone & Joint, Charlotte, North Carolina
  - Rheumatology, Durham, North Carolina
  - Physicians East, Pa, Greenville, North Carolina
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Center For Arthritis Therapy And Research, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Pro Research, Eugene, Oregon
  - Portland Rheumatology Clinic, Llc, Lake Oswego, Oregon
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Rheumatology Associates, Providence, Rhode Island
  - Low Country Rheumatology, Pa, Charleston, South Carolina
  - Columbia Arthritis Center, Columbia, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Acme Research, Llc, Orangeburg, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - Rheumatology Consultants Pllc, Knoxville, Tennessee
  - The Arthritis Group, Pc, Memphis, Tennessee
  - St. Thomas Hospital Tower East, Nashville, Tennessee
  - Walter F. Chase, Austin, Texas
  - Rheumatic Disease Clinical Research Center, Llc, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Texas Research Center, Sugarland, Texas
  - Arthritis Clinic Of Northern Virginia, P.C., Arlington, Virginia
  - Center For Arthritis & Rheumatic Diseases, Pc, Chesapeake, Virginia
  - South Puget Sound Clinincal Research Center, Olympia, Washington
  - Tacoma Center For Arthritis Research Ps, Tacoma, Washington
- Argentina (6):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad Autonoma, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe, Santa Fe Province
  - Local Institution, Santa Fe, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Australia (6):
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Cairns, Queensland
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Woodville, South Australia
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Shenton Park, Western Australia
- Belgium (5):
  - Local Institution, Brussels
  - Local Institution, Hasselt
  - Local Institution, Leuven
  - Local Institution, Wilrijk
  - Local Institution, Yvoir
- Brazil (8):
  - Local Institution, Goiânia, Goiás
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Recife, Pernambuco
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (8):
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Hamilton, Ontario
  - Local Institution, Mississauga, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Trois-Rivières, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Santiago, Santiago Metropolitan, Chile
- France (10):
  - Local Institution, Bordeaux
  - Local Institution, Brest
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Le Mans
  - Local Institution, Lille
  - Local Institution, Marseille
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Leipzig
  - Local Institution, München
- Local Institution, Heraklion Crete, Greece
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Debrecen
- India (7):
  - Local Institution, Secunderabad, Andhra Pradesh
  - Local Institution, Navrangpura, Ahmedabad, Gujarat
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Bangalore
  - Local Institution, Hyderabad
  - Local Institution, Lucknow
  - Local Institution, New Delhi
- Local Institution, Dublin, Dublin, Ireland
- Italy (5):
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Pavia
  - Local Institution, Roma
  - Local Institution, Siena
- Mexico (10):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Nuevo León, Nuevo León
  - Local Institution, Querétaro City, Querétaro
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Mérida, Yucatán
- Local Institution, Leeuwarden, Netherlands
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Callao, Provincia Constitucional del Callao
- Poland (7):
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Gmina Końskie
  - Local Institution, Krakow
  - Local Institution, Poznan
  - Local Institution, Torun
  - Local Institution, Warsaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Yaroslavl
  - Local Institution, Yekaterinburg
- South Africa (5):
  - Local Institution, Kempton Park, Gauteng
  - Local Institution, Muckleneuk, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
- South Korea (4):
  - Local Institution, Seoul, Sungdong-Gu
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Seoul
- Taiwan (2):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
- Turkey (Türkiye) (3):
  - Local Institution, Denizli
  - Local Institution, Edirne
  - Local Institution, Gaziantep
- United Kingdom (5):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, Bridgend, Glamorgan
  - Local Institution, London, Greater London
  - Local Institution, Southampton, Hampshire
  - Local Institution, Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- [Derived] Alten R, Bingham CO 3rd, Cohen SB, Curtis JR, Kelly S, Wong D, Genovese MC. Antibody response to pneumococcal and influenza vaccination in patients with rheumatoid arthritis receiving abatacept. BMC Musculoskelet Disord. 2016 May 26;17:231. doi: 10.1186/s12891-016-1082-z. PMID 27229685
- [Derived] Genovese MC, Tena CP, Covarrubias A, Leon G, Mysler E, Keiserman M, Valente R, Nash P, Simon-Campos JA, Box J, Legerton CW 3rd, Nasonov E, Durez P, Delaet I, Teng J, Alten R. Subcutaneous abatacept for the treatment of rheumatoid arthritis: longterm data from the ACQUIRE trial. J Rheumatol. 2014 Apr;41(4):629-39. doi: 10.3899/jrheum.130112. Epub 2014 Mar 1. PMID 24584926
- [Derived] Genovese MC, Covarrubias A, Leon G, Mysler E, Keiserman M, Valente R, Nash P, Simon-Campos JA, Porawska W, Box J, Legerton C 3rd, Nasonov E, Durez P, Aranda R, Pappu R, Delaet I, Teng J, Alten R. Subcutaneous abatacept versus intravenous abatacept: a phase IIIb noninferiority study in patients with an inadequate response to methotrexate. Arthritis Rheum. 2011 Oct;63(10):2854-64. doi: 10.1002/art.30463. PMID 21618201
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the double blind short term (ST) period of the Main study, a sub-study in RA participants was initiated to evaluate anti-tumor necrosis factor (TNF) failure population. The sub-study was terminated early due to slow recruitment and participants from the sub-study were allowed to roll into the Main study during the LT Open Label Period.
Pre-assignment Details: 2492 enrolled: 2472 in Main Study:1008 not randomized: 918 no longer met criteria, 61 withdrew consent, 7 lost to follow-up, 22 other reasons. Randomized, not treated: 4 no longer met criteria, 2 withdrew consent, and 1 randomization error; 20 enrolled in Anti-TNF sub-study; 2 not randomized as no longer met criteria; 18 randomized in substudy.
Groups:
- Subcutaneous (SC) Abatacept: During the Main Study Double Blind ST Period, participants received 125 mg weekly SC abatacept injections for 6 months (with an IV abatacept loading dose on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV Placebo) with the exception that on Day 1 a loading dose of IV abatacept replaced the IV Placebo treatment. During the Open Label Long Term (LT) Period, participants in both the Main Study and the Anti-TNF Failure Sub-study switched to open-label SC abatacept. The study continued until SC formulation became commercially available on a country basis or the Sponsor terminated the study.
- Intravenous (IV) Abatacept: During the Main study Double Blind ST Period, participants received IV abatacept infusions on Days 1, 15, 29, and every 28 days, thereafter for 6 months. A double-dummy design was used to protect the blind, thus, participants also received SC injections of placebo (SC Placebo). During the Open Label LT Period, participants in both the Main Study and the Anti-TNF Failure Sub-study switched to open-label SC abatacept. The study continued until SC formulation became commercially available on a country basis or the Sponsor terminated the study.
Period: Double Blind ST Period Main Study
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept
Started | 736 (Randomized and treated) | 721 (Randomized and treated)
Completed | 693 | 676
Not Completed | 43 | 45
Not completed — Adverse Event | 17 | 25
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Lost to Follow-up | 0 | 6
Not completed — Administrative Reason By Sponsor | 1 | 0
Not completed — Death | 1 | 1
Not completed — No Longer Meets Study Criteria | 2 | 1
Not completed — Lack of Efficacy | 6 | 1
Not completed — Poor/Non-Compliance | 3 | 0
Not completed — Missed Doses | 0 | 1
Not completed — Incomplete Breast Exam | 0 | 1
Not completed — Suspended Drug Due To Surgery | 0 | 1
Not completed — Early Discontinuation | 0 | 1
Not completed — Participant Weight Gain | 1 | 0
Not completed — Participant Withdrew-Recurrent Infection | 0 | 1
Not completed — Investigator Decision | 0 | 1
Not completed — Ongoing Infection Risk | 1 | 0
Period: Anti-TNF Sub-Study in ST Period
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept
Started | 8 (7 completed Sub-Study ST period and 6 chose to roll over into LT Period.) | 10 (9 completed Sub-Study ST Period and 9 chose to over into the LT Period.)
Completed | 7 | 9
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Period: Open Label LT Period Main + Sub-Study
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept
Started | 1373 (1373 includes 15 participants from ST Period Sub-Study who rolled over into LT Period (6 SC + 9 IV).) | 0 (IV administration was discontinued and abatacept was only administered SC during LT Period.)
Completed | 945 | 0
Not Completed | 428 | 0
Not completed — Adverse Event | 100 | 0
Not completed — Withdrawal by Subject | 81 | 0
Not completed — Pregnancy | 16 | 0
Not completed — Lost to Follow-up | 32 | 0
Not completed — Administrative reason by Sponsor | 9 | 0
Not completed — Death | 20 | 0
Not completed — No longer met criteria | 1 | 0
Not completed — Lack of Efficacy | 89 | 0
Not completed — Poor/non-compliance | 8 | 0
Not completed — non-specified | 71 | 0
Not completed — no end of study status page | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per-protocol Population in ST Period.
Groups:
- Subcutaneous (SC) Abatacept: Participants received 125 mg weekly SC abatacept injections (with an intravenous [IV] abatacept loading dose on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV Placebo) with the exception that on Day 1 a loading dose of IV abatacept replaced the IV Placebo treatment. The Per Protocol (PP) Analysis Population (instead of the Intent-To-Treat Population) was used to perform primary and key secondary efficacy analyses as per regulatory guidelines for non-inferiority studies.
- Intravenous (IV) Abatacept: Participants received IV abatacept infusions on Days 1, 15, 29, and every 28 days, thereafter. A double-dummy design was used to protect the blind, thus, participants also received SC injections of placebo (SC Placebo). The Per Protocol (PP) Analysis Population (instead of the Intent-To-Treat Population) was used to perform primary and key secondary efficacy analyses as per regulatory guidelines for non-inferiority studies.
- Total: Total of all reporting groups
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept | Total
Number analyzed (Participants) | 696 | 683 | 1379
Age, Continuous [Mean (Standard Deviation); unit: years] — Since regulatory guidelines indicate use of the Per Protocol (PP) Analysis Population (instead of the Intent-To-Treat Population) for non-inferiority studies, this population was used to perform primary and key secondary efficacy analyses. Thus, Baseline continuous age data are presented for the PP Analysis Population.
  years | 49.9 (13.0) | 49.9 (12.7) | 49.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 586 | 549 | 1135
  Male | 110 | 134 | 244
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 63 | 72 | 135
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 24 | 50
  White | 516 | 505 | 1021
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 86 | 81 | 167
Region Of Enrollment [Number; unit: participants]
  North America | 129 | 111 | 240
  South America | 338 | 340 | 678
  Europe | 123 | 123 | 246
  Rest of the World | 106 | 109 | 215
Baseline Weight Category [Number; unit: participants]
  <60 kg | 175 | 171 | 346
  60 to 100 kg | 464 | 465 | 929
  >100 kg | 57 | 47 | 104
Duration of RA Disease [Mean (Standard Deviation); unit: years] | 7.6 (8.0) | 7.7 (7.9) | 7.7 (7.9)
Duration of Disease Category [Number; unit: participants]
  ≤2 Years | 229 | 206 | 435
  2 - ≤5 yrs | 144 | 145 | 289
  5 - ≤10 yrs | 134 | 155 | 289
  > 10 yrs | 189 | 177 | 366
Number of Tender Joints [Mean (Standard Deviation); unit: tender joints] — Tender joints are an indicator of Rheumatoid Arthritis. The number of tender joints in a standard 68 joint count was evaluated. The number of tender joints ranges from 0 tender joints to 68, where an increased number of tender joints indicates increasing level of disease severity.
  tender joints | 30 (14.1) | 29.2 (13.1) | 29.6 (13.6)
Number of Swollen Joints [Mean (Standard Deviation); unit: swollen joints] — Swollen joints are an indicator of Rheumatoid Arthritis. The number of swollen joints in a standard 66 joint count was evaluated. The number of swollen joints ranges from 0 swollen joints to 66, where an increased number of swollen joints indicates increasing level of disease severity.
  swollen joints | 20.5 (9.4) | 19.6 (8.5) | 20.0 (9.0)
Participant Pain Assessment [Mean (Standard Deviation); unit: units on a scale] — The participant self-reported pain assessment is a core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale (VAS) with 0 mm representing no pain and 100 mm representing the most pain possible. For each post-baseline visit in the DB, time-matched baseline Participant Pain Assessment values were presented and represent the mean baseline value for only that cohort of participants with assessments available at that visit.
  units on a scale | 68.0 (20.0) | 66.9 (20.5) | 67.5 (20.3)
Physical Function (Health Assessment Questionnaire Disability Index [HAQ-DI]) [Mean (Standard Deviation); unit: units on a scale] — The disability section of the full HAQ includes 20 questions to assess physical The HAQ-DI includes 20 questions to assess physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do. HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. HAQ-DI overall score ranges from a minimum of 0 to a maximum of 3.0.
  units on a scale | 1.73 (0.68) | 1.69 (0.67) | 1.71 (0.67)
Participant Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Participants used a horizontal VAS of 100 mm for overall assessment of rheumatoid arthritis. Scale ranged from 0 (very well) to 100 (very poor). Participants were instructed to draw a vertical through a horizontal line to indicate state of rheumatoid arthritis. Distance from the "very well" end of the horizontal line to the vertical line drawn by the participant was the global disease assessment score on a scale of 1-10, where 1=controlled or equivocal rheumatoid arthritis activity, 1.1-4=mild activity, 4-8=moderate activity, and 8.1-10=high activity.
  units on a scale | 67.2 (20.1) | 65.2 (19.9) | 66.2 (20.0)
Physician Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Physician global rheumatoid arthritis assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale, with 0 mm representing no pain and 100 mm representing the most pain possible.
  units on a scale | 64.3 (16.5) | 63.4 (16.3) | 63.9 (16.4)
High Sensitivity C-Reactive Protein (hsCRP) Level [Mean (Standard Deviation); unit: mg/dL] — hs-CRP is a acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). Levels of hs-CRP can be used to determine DAS28.
  mg/dL | 2.65 (2.91) | 2.72 (2.91) | 2.69 (2.91)
Disease Activity Score (CRP) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 index measures disease activity in rheumatoid arthritis and is a composite derived from the number of swollen/tender joints, laboratory tests of inflammation (C-reactive protein measured in mg/L), and participant assessment of global health (by marking a 100 mm line from "very good" to "very bad"). A higher DAS28 score indicates worse control of disease. High disease activity is > 5.1, low disease activity is < 3.2 and remission is < 2.6.
  units on a scale | 6.25 (0.84) | 6.22 (0.83) | 6.24 (0.83)
Rheumatoid Factor Status [Number; unit: participants] — Rheumatoid factor (RF or RhF) is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process. A positive value for RF was >20 IU/mL; a negative value for RF was ≤ 20 IU/mL.
  participants
    Negative | 102 | 91 | 193
    Positive | 582 | 583 | 1165
    Unknown | 12 | 9 | 21
Baseline Methotrexate (MTX) Dose [Mean (Standard Deviation); unit: mg/wk] | 16.3 (3.6) | 16.5 (3.7) | 16.4 (3.6)
Weight [Mean (Standard Deviation); unit: kg] | 72.1 (18.1) | 71.5 (17.5) | 71.8 (17.8)

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Period: Number of Participants Achieving American College of Rheumatology (ACR) 20 Response at Day 169
Description: The ACR 20 definition of improvement is a 20% improvement from baseline in the number of tender and swollen joints, and a 20% improvement from baseline in 3 of the remaining 5 core set measures: participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function and acute phase reactant value (C-reactive protein).
Time Frame: Day 169
Population: Per protocol (PP) population, defined as participants who are compliant with the study criteria.
Measure: Number; unit: participants
Groups:
- Subcutaneous Abatacept: Participants received weekly injections of 125 mg subcutaneous abatacept (with a loading dose of intravenous (IV) abatacept on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV placebo) with the exception that on Day 1, a loading dose of IV abatacept replaced the IV placebo treatment.
- Intravenous Abatacept: Participants received IV abatacept infusions on Days 1, 15, and 29 and every 28 days thereafter. A double-dummy design was used to protect the blind, thus, participants also received subcutaneous injections of placebo (subcutaneous placebo).
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 693 | 678
participants | 527 | 514

2. Secondary Outcome: Double-blind Period: Number of Participants Achieving ACR 50 and ACR 70 Responses at Day 169
Description: The ACR 50 definition of improvement is a 50% improvement from baseline in the number of tender and swollen joint counts, and a 50% improvement from baseline in 3 of the remaining 5 core set measures: participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function and acute phase reactant value (C-reactive protein). ACR 70 is defined similarly with 70% improvements from baseline for tender and swollen joint counts and 3 out of 5 core measures.
Time Frame: Day 169
Population: PP population, defined as participants who are compliant with the study criteria.
Measure: Number; unit: participants
Groups:
- Subcutaneous Abatacept: Participants received weekly injections of 125 mg subcutaneous abatacept (with a loading dose of IV abatacept on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV placebo) with the exception that on Day 1, a loading dose of IV abatacept replaced the IV placebo treatment.
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 693 | 678
participants
  ACR 50 | 357 | 341
  ACR 70 | 183 | 170

3. Secondary Outcome: Double-blind Period: Mean Baseline Health Assessment Questionnaire Disability Index (HAQ-DI) for Participants With Assessments at Day 169
Description: The disability section of the full HAQ-DI includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. Higher scores=greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered.
Time Frame: Day 169
Population: All participants who received at least 1 dose of study medication at any time and had HAD-QI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 729 | 711
units on a scale | 1.72 (0.68) | 1.67 (0.67)

4. Secondary Outcome: Double-blind Period: Adjusted Mean Change From Baseline to Day 169 in HAQ-DI
Description: The HAQ-DI includes 20 questions to assess physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do. HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. HAQ-DI ranges from 0 to a maximum overall score of 3.0.
Time Frame: Baseline to Day 169
Population: All participants who received at least 1 dose of study medication at any time and had HAD-QI scores available.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Intravenous Abatacept: Participants received IV abatacept infusions on Days 1, 15, and 29 and every 28 days thereafter. A double-dummy design was used to protect the blind, thus, participants also received subcutaneous injections of placebo (Subcutaneous placebo placebo).
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 729 | 711
units on a scale | -0.69 (0.02) | -0.70 (0.02)

5. Secondary Outcome: Double-blind Period: Number of Participants Achieving Clinically Meaningful HAQ-DI Response at Day 169
Description: The disability section of the full HAQ-DI includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3=unable to do. Higher scores=greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ-DI response=an improvement of at least 0.3 units from baseline in HAQ-DI.
Time Frame: Day 169
Population: All participants who received at least 1 dose of study medication at any time and had HAD-QI scores available
Measure: Number; unit: participants
Groups:
- Subcutaneous Abatacept: Participants received weekly injections of 125 mg subcutaneous abatacept (with an IV abatacept loading dose on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV Placebo) with the exception that on Day 1 a loading dose of IV abatacept replaced the IV Placebo treatment.
- Intravenous Abatacept: Participants received IV abatacept infusions on Days 1, 15, 29, and every 28 days, thereafter. A double-dummy design was used to protect the blind, thus, participants also received SC injections of placebo (SC Placebo).
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 729 | 711
participants | 483 | 442

6. Secondary Outcome: Double-blind Period: Number of Participants With Death As Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Treatment-related AEs, or AEs Leading to Discontinuation
Description: AE=any new untoward medical event or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Treatment-related SAE=possibly, probably, or certainly related to study drug
Time Frame: Day 1 to 56 days after last dose in short-term or first dose in the long-term, whichever occurs first.
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Subcutaneous Abatacept: Participants received weekly injections of 125 mg subcutaneous abatacept (with a loading dose of IV abatacept on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV placebo) with the exception
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants
  Deaths | 2 | 5
  SAEs | 31 | 35
  Treatment-related SAEs | 5 | 12
  SAEs Leading to Discontinuation | 8 | 14
  AEs | 493 | 470
  Treatment-related AEs | 204 | 210
  AEs Leading to Discontinuation | 15 | 25

7. Secondary Outcome: Anti-TNF Failure Sub-study Double-blind Period: Number of Participants With SAEs, AEs Leading to Discontinuation or Who Died
Description: AE=any new untoward medical event or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: Day 1 to 56 days after last dose in short-term or first dose in the long-term, whichever occurs first.
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Subcutaneous (SC) Abatacept: During the Double Blind ST Period, participants received 125 mg weekly SC abatacept injections for 6 months (with an intravenous [IV] abatacept loading dose on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV Placebo) with the exception that on Day 1 a loading dose of IV abatacept replaced the IV Placebo treatment. An Anti-TNF Failure Sub-study was initiated using the same treatment as the Main study in order to assess the immunogenicity and safety in the Anti-TNF Failure population.
- Intravenous (IV) Abatacept: During the Double Blind ST Period, participants received IV abatacept infusions on Days 1, 15, 29, and every 28 days, thereafter for 6 months. A double-dummy design was used to protect the blind, thus, participants also received SC injections of placebo (SC Placebo). An Anti-TNF Failure Sub-study was initiated using the same treatment as the Main study in order to assess the immunogenicity and safety in the Anti-TNF Failure population.
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept
Number analyzed (Participants) | 8 | 10
participants
  Deaths | 0 | 0
  SAEs | 0 | 0
  AEs Leading to Discontinuation | 0 | 0

8. Secondary Outcome: Double-blind Period: Number of Participants With AEs of Special Interest
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs: all infections,serious infections,and opportunistic infections; autoimmune disorders; malignancies; acute infusional AEs (prespecified AEs occurring within 1 hr of start of infusion), peri-infusional AEs (prespecified AEs occurring within 24 hrs of the start of infusion), system injection reactions, and local injection site reactions
Time Frame: Day 1 up to 56 days post last dose in short- term period or first dose in the long -term period, whichever occurs first.
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants
  Infections | 234 | 221
  Malignancies | 3 | 5
  Autoimmune Disorders | 7 | 6
  Acute Infusional AEs | 20 | 16
  Peri-infusional AEs | 59 | 59
  Local Injection Site Reactions | 19 | 18
  Systemic Injection Reactions | 56 | 56

9. Secondary Outcome: Double-blind Period: Number of Participants With Clinically Significant Abnormalities in Vital Sign Measurements
Description: Vital sign measurements were performed for participants before and after infusion/subcutaneous injection of study medication at each visit and included seated systolic blood pressure, seated diastolic blood pressure, temperature, and heart rate. Abnormalities were determined to be clinically significant by the investigator.
Time Frame: Day 1 through end of short-term period (Day 169)
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Intravenous Abatacept: Participants received weekly injections of 125 mg subcutaneous abatacept (with a loading dose of IV abatacept on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV placebo) with the exception that on Day 1, a loading dose of IV abatacept replaced the IV placebo treatment.
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants | 0 | 0

10. Secondary Outcome: Double-blind Period: Number of Participants With Hematology Laboratory Test Results Meeting the Criteria for Marked Abnormality
Description: ULN=upper limit of normal; LLN=lower limit of normal; BL= baseline. Marked abnormality criteria: Hemoglobin: >3 g/dL decrease from BL; hematocrit: <0.75*BL; erythrocytes: <0.75*BL; platelets: <0.67*LLN/>1.5*ULN, or if BL<LLN, use <0.5*BL and <100,000 mm^3; leukocytes: <0.75*LLN/>1.25*ULN, or if BL<LLN use <0.8*BL or >ULN, or if BL>ULN, use >1.2*BL or <LLN; neutrophils+bands: <1.0*10^3 c/uL; eosinophils: >0.750*10^3 c/uL; basophils: >400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750*10^3 c/uL/>7.50*10^3 c/uL.
Time Frame: Day 1 through end of short-term period (Day 169)
Population: All randomized participants who received at least 1 dose of study medication. n=Number of participants with assessments available.
Measure: Number; unit: participants
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants
  Low hemoglobin (LLN=11.5 g/dL); n=729, 713 | 2 | 5
  Low hematocrit (LLN=34%); n=726, 713 | 2 | 4
  Low erythrocytes(LLN=3.8 x10*6c/uL);n=729, 713 | 2 | 3
  Low platelets (LLN=140*10^9 c/L); n=725, 709 | 1 | 0
  High platelets (ULN=450*10^9 c/L); n=725, 709 | 0 | 0
  Low leukocytes (LLN= 3.8*10^3 c/uL); n=729, 713 | 6 | 2
  High leukocytes (ULN = 10.6*10^3 c/uL);n=729, 713 | 25 | 18
  Low neutrophils+bands(LLN=1.8*10^3 c/uL);n=730,713 | 0 | 0
  High eosinophils (ULN= 7*10^3 c/uL); n=730, 712 | 22 | 16
  High basophils (ULN= 0.2*10^3 c/uL); n=730, 712 | 0 | 0
  High monocytes (ULN=1*10^3 c/uL); n=730, 712 | 0 | 1
  Low lymphocytes (LLN= 0.7*10^3 c/uL);n=730,712 | 40 | 42
  High lymphocytes(ULN=4.5*10^3 c/uL);n=730,712 | 40 | 42

11. Secondary Outcome: Double-blind Period: Number of Participants With Liver Function Laboratory Test Results Meeting the Criteria for Marked Abnormality
Description: Marked abnormality criteria: Alkaline phosphatase (ALP): >2*ULN, or if BL>ULN, use >3*BL; aspartate aminotransferase (AST): >3*ULN, or if BL>ULN, use >4*BL; alanine aminotransferase (ALT): >3*ULN, or if BL>ULN, use >4*BL; G-glutamyl transferase (GGT): >2* ULN, or if BL>ULN, use >3*BL; bilirubin: >2* ULN, or if BL>ULN, use >4*BL; blood urea nitrogen: >2* BL; creatinine: >1.5*BL
Time Frame: Day 1 through end of short-term period (Day 169)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants
  High ALP (ULN=400 U/L); n=730, 713 | 1 | 3
  High AST (ULN=44 U/L); n=729, 713 | 5 | 5
  High ALT (ULN=55 U/L);n=729, 713 | 12 | 16
  High GGT (ULN=65 U/L); n=730, 713 | 8 | 14
  High bilirubin (ULN=1.2 mg/dL); n=730, 713 | 1 | 0
  High blood urea nitrogen (26 mg/dL); n=730, 713 | 21 | 27
  High creatinine (ULN=1.5 mg/dL); n=730, 713 | 19 | 30

12. Secondary Outcome: Double-blind Period: Number of Participants With Electrolyte Laboratory Test Results Meeting the Criteria for Marked Abnormality
Description: Marked abnormality criteria: Sodium: <0.95*LLN/>1.05*ULN, or if BL<LLN, use <0.95* BL or >ULN, or if BL>ULN, use>1.05* BL or <LLN; potassium: <0.9* LLN/>1.1*ULN, or if BL<LLN then use <0.9* BL or >ULN, or if BL>ULN, use>1.1* BL or <LLN; chlorine: <0.9*LLN/>1.1* ULN, or if BL<LLN, use <0.9*BL or >ULN, or if BL>ULN, use>1.1*BL or <LLN; calcium: <0.8* LLN/>1.2* ULN, or if BL<LLN, use <0.75*BL or >ULN, or if BL>ULN, use>1.25* BL or <LLN; phosphorous: <0.75* LLN/>1.25*ULN, or if BL<LLN, use 0.67*BL or >ULN, or if BL>ULN, use>1.33* BL or <LLN
Time Frame: Day 1 through end of short-term period (Day 169)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants
  Low sodium (LLN=135 mEq/L) | 2 | 0
  High sodium (ULN=148 mEq/L) | 0 | 0
  Low potassium (LLN=3.5 mEq/L) | 9 | 9
  High potassium (ULN=5.5 mEq/L) | 1 | 0
  Low chlorine (LLN= 96 mEq/L) | 0 | 0
  High chlorine (ULN=109 mEq/L) | 0 | 0
  Low calcium (LLN=8.4 mg/dL) | 1 | 0
  High calcium (ULN=10.6 mg/dL) | 1 | 0
  Low phosphorous (LLN=0.8 mg/dL) | 1 | 2
  High phosphorous (ULN=5.6 mg/dL) | 0 | 1

13. Secondary Outcome: Double-blind Period: Minimum Observed Serum Concentration of Abatacept
Time Frame: Days 57, 85, 113, 120, 127, 134, 141, and 169
Population: Participants who received at least 1 dose of study medication and from whom at least 1 pharmacokinetic (PK) sample was collected and reported (N). Only participants with adequate PK profiles were included in the summary statistics and statistical analysis (n).
Measure: Geometric Mean (Standard Deviation); unit: µg/mL
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 630 | 649
µg/mL
  Day 57 (n=25, n=16) | 31.60 (21.483) | 23.14 (14.008)
  Day 85 (n=630, n=649) | 28.30 (21.692) | 20.00 (13.441)
  Day 113 (n=44, n=29) | 26.49 (16.569) | 18.76 (16.322)
  Day 120 (n=27) | 25.10 (14.933) | NA (NA) — PK values were not sampled for IV abatacept group on Day 120
  Day 127 (n=28) | 29.16 (14.780) | NA (NA) — PK values were not sampled for IV abatacept group on Day 127
  Day 134 (n=27) | 25.10 (15.753) | NA (NA) — PK values were not sampled for IV abatacept group on Day 134
  Day 141 (n=26, n=26) | 25.79 (14.264) | 18.10 (17.717)
  Day 169 (n=530, n=521) | 24.91 (14.989) | 18.10 (17.94)

14. Secondary Outcome: Anti-TNF Failure Sub-study Double-blind Period: Minimum Observed Serum Concentration (Cmin) of Abatacept
Description: Serum concentrations of abatacept were analyzed using a validated ELISA. Steady-state trough observed concentration in serum (Cminss) was measured in μg/mL. Samples were obtained on Days 57, 85, 113, 120, 127, 134, 141, and 169.
Time Frame: Days 57, 85, 113, 120, 127, 134, 141, and 169 (ST Period)
Population: Participants who received at least 1 dose of study medication and who had adequate PK profiles were analyzed. n= number of participants available at each specific time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept
Number analyzed (Participants) | 6 | 9
μg/mL
  Day 57 (n=3,4) | 25.53 (16) | 15.51 (25)
  Day 85 (n=6,9) | 21.51 (26) | 12.50 (48)
  Day 113 (n=6,6) | 23.14 (27) | 11.10 (31)
  Day 120 (n=4) | 25.75 (17) | NA (NA) — PK values were not sampled for IV abatacept group on Day 120.
  Day 127 (n=3) | 25.42 (9) | NA (NA) — PK values were not sampled for IV abatacept group on Day 127.
  Day 134 (n=3) | 25.55 (13) | NA (NA) — PK values were not sampled for IV abatacept group on Day 134.
  Day 141 (n=4,6) | 20.85 (24) | 8.34 (44)
  Day 169 (n=5,7) | 19.66 (25) | 9.00 (53)

15. Secondary Outcome: Double-blind Period: Maximum Observed Serum Concentration of Abatacept
Time Frame: End of infusion on Days 1 and 113 for IV infusion and in the dosing interval of Days 113 to 120 for subcutaneous
Population: Participants who received at least 1 dose of study medication and who had adequate PK profiles for analysis
Measure: Geometric Mean (Standard Deviation); unit: µg/mL
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 39 | 39
µg/mL | 40.39 (30.148) | 222.35 (71.920)

16. Secondary Outcome: Anti-TNF Failure Substudy Double Blind Period: Geometric Mean Maximum Observed Serum Concentration of Abatacept
Description: Serum concentrations of abatacept were analyzed using a validated enzyme-linked immunosorbent assay (ELISA). Samples were obtained on Days 57, 85, 113, 120, 127, 134, 141, and 169. Cmax was measured in micrograms per milliliter (μg/mL).
Time Frame: End of infusion on Days 1 and 113 for IV infusion and in the dosing interval of Days 113 to 120 for subcutaneous
Population: Participants in the Sub-study who received at least 1 dose of study medication and who had adequate PK profiles were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept
Number analyzed (Participants) | 5 | 5
μg/mL | 35.84 (24) | 229.88 (26)

17. Secondary Outcome: Double-blind Period: Area Under The Curve In A Dose Interval (AUC TAU) of Abatacept
Time Frame: Dosing interval between Days 113 and 141 (TAU=28 days)
Population: Participants who received at least 1 dose of study medication and who had adequate PK profiles for analysis
Measure: Geometric Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 39 | 39
µg*h/mL | 5182.37 (2854.136) | 39587.08 (15444.743)

18. Secondary Outcome: Anti-TNF Failure Sub-study Double Blind Period: Area Under The Curve In A Dose Interval (AUC TAU) of Abatacept
Description: Serum concentrations of abatacept were analyzed using a validated ELISA. AUC(TAU) was measured as μg*h/mL. Samples for AUC (TAU) were obtained on Days 113, 120, 127, 134, and 141.
Time Frame: Dosing Interval between Days 113 and 141 (TAU=28 days)
Population: Participants in the sub-study who received at least 1 dose of study medication and who had adequate PK profiles for analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Subcutaneous (SC) Abatacept | Intravenous (IV) Abatacept
Number analyzed (Participants) | 5 | 6
μg*h/mL | 4384.80 (17) | 34260.55 (35)

19. Secondary Outcome: Double-blind Period: Number of Participants With Positive Anti-abatacept or Anti-Cytotoxic T Lymphocyte Antigen 4-T Cell (CTLA4-T) Responses Over Time by Enzyme Linked Immunoabsorbant Assay (ELISA)
Description: Serum samples from all treated adult participants with active rheumatoid arthritis were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept (anti-ABA) or anti-CTLA4 antibody (anti-CTLA4).
Time Frame: Days 85, and 169 and postvisits on Days 28, 56, and 85
Population: All randomized participants who received at least 1 dose of study medication. n=Number of participants with at least 1 assessment available.
Measure: Number; unit: participants
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants
  Day 85 anti-ABA (n=700, n=682) | 0 | 2
  Day 85 anti-CTLA4 (n=705, n=689 | 0 | 0
  Day 85 total (n=706, n=689) | 0 | 2
  Day 169 anti-ABA (n=671, n=648) | 3 | 4
  Day 169 anti-CTLA4 (n=681, n=658) | 2 | 4
  Day 169 total (n=681, n=658) | 5 | 8
  Overall on-treatment visits anti-ABA (n=707, 691) | 3 | 5
  Overall on-treatment visits anti-CTLA4 (n=716,702) | 2 | 4
  Overall on-treatment visits total (n=716, 702) | 5 | 9
  28 days post last dose anti-ABA (n=18, n=25) | 0 | 0
  28 days post last dose anti-CTLA4 (n=20, n=27) | 0 | 2
  28 days post last dose total (n=20, n=27) | 0 | 2
  56 days post last dose anti-ABA (n=19, n=22) | 0 | 0
  56 days post last dose anti-CTLA4 (n=19, n=23) | 1 | 1
  56 days post last dose total (n=19, n=23) | 1 | 1
  85 days post last dose anti-ABA (n=12, n=15) | 0 | 0
  85 days post last dose anti-CTLA4 (n=13, n=15) | 2 | 5
  85 days post last dose total (n=13, n=15) | 2 | 5
  Overall post visits anti-ABA (n=26, n=29) | 0 | 0
  Overall post visits anti-CTLA4 (n=28, n=31) | 3 | 7
  Overall post visits total (n=28, n=31) | 3 | 7
  Overall anti-ABA (n=714, n=698) | 3 | 5
  Overall anti-CTLA4 (n=725, n=710) | 5 | 11
  Overall total (n=725, n=710) | 8 | 16

20. Secondary Outcome: Double-blind Period: Time-matched Median Percent Change From Baseline in Levels of Serum C-reactive Protein Over the Short-term Period
Description: C-reactive protein is an acute phase reactant protein that is a clinical marker for rheumatoid arthritis. Time-matched median percent change from baseline= (time-matched baseline value - Post-baseline value)/time-matched baseline value*100, where the time-matched baseline value represents the median baseline value for only that cohort of participants with measurements available at that visit.
Time Frame: Baseline to Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
percent change
  Day 15 (n=720, n=703) | 34.16 [-11.11 to 58.80] | 33.74 [-6.24 to 58.41]
  Day 29 (n=727, n=711) | 39.74 [3.83 to 66.99] | 42.52 [0.42 to 68.66]
  Day 57 (n=727, n=711) | 47.88 [6.84 to 73.53] | 51.42 [7.53 to 74.95]
  Day 85 (n=727, n=711) | 52.90 [8.70 to 78.25] | 53.65 [11.05 to 79.42]
  Day 113 (n=727, n=711) | 53.33 [7.09 to 80.29] | 58.12 [11.21 to 81.26]
  Day 141 (n=727, n=711) | 56.12 [5.28 to 83.24] | 58.39 [16.14 to 81.52]
  Day 169 (n=727, n=711) | 57.18 [11.18 to 83.28] | 56.81 [17.92 to 82.70]

21. Secondary Outcome: Double-blind Period: Number of Participants With Positive Anti-abatacept Responses Over Time by Electrochemiluminescence Immunoassay Among the First 10% of Participants Randomized
Description: An electrochemiluminescence immunoassay screened sera for drug-specific antibodies, immunocompetition was used to identify specific anti-abatacept reactivity. CTLA4 and Possibly Ig category=reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; abatacept molecule). Ig and/or Junction (JNCT) category=reactivity against constant regions and/or hinge region of human IgG1. Drug-induced seropositivity was defined as a postbaseline titer higher than Baseline, or any postbaseline positivity if Baseline value was missing. Trt=treatment.
Time Frame: Days 85, and 169 and postvisits on Days 28, 56, and 85
Population: All participants who received at least 1 dose of abatacept and had at least 1 immunogenicity result reported during the short-term period.
Measure: Number; unit: participants
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 82 | 71
participants
  Day 85 CTLA4 + possibly Ig (n=78, n=67) | 0 | 0
  Day 85 Ig +/- JNCT (n=78, n=67) | 0 | 0
  Day 85 total (n=78, n=67) | 0 | 0
  Day 169 CTLA4 + possibly Ig (n=75, n=67) | 0 | 1
  Day 169 Ig +/- JNCT (n=75, n=67) | 0 | 0
  Day 169 total (n=75, n=67) | 0 | 1
  Overall on-TRT CTLA4 + possibly Ig (n=79, 70) | 0 | 1
  Overall on-TRT Ig +/- JNCT (n=79, 70) | 0 | 0
  Overall on-TRT total (n=79, 70) | 0 | 1
  28 days post last dose CTLA4+possibly Ig (n=2,n=2) | 0 | 0
  28 days post last dose Ig +/- JNCT (n=2, n=2) | 0 | 0
  28 days post last dose Total (n=2, n=2) | 0 | 0
  56 days post last dose CTLA4+possibly Ig (n=2,n=2) | 0 | 0
  56 days post last dose Ig +/- JNCT (n=2, n=2) | 0 | 0
  56 days post last dose total (n=2, n=2) | 0 | 0
  85 days post last dose CTLA4+possibly Ig (n=1,n=1) | 0 | 0
  85 days post last dose Ig +/- JNCT (n=1, n=1) | 0 | 0
  85 days post last dose total (n=1, n=1) | 0 | 0
  Overall post visits CTLA4+possibly Ig (n=3, n=2) | 0 | 0
  Overall post visits Ig +/- JNCT (n=3, n=2) | 0 | 0
  Overall post visits total (n=3, n=2) | 0 | 0
  Overall CTLA4+possibly Ig (n=82, n=71) | 0 | 1
  Overall Ig +/- JNCT (n=82, n=71) | 0 | 0
  Overall total (n=82, n=71) | 0 | 1

22. Secondary Outcome: Double-blind Period: Number of Participants Seroconverting by Day 169 According to Status (Negative or Positive) at Baseline
Description: Rheumatoid factor (RF) is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process.
Time Frame: Baseline to Day 169
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 736 | 721
participants
  Baseline RF negative | 106 | 93
  Baseline RF negative; Day 169 RF positive | 2 | 3
  Baseline RF positive | 586 | 582
  Baseline RF positive ; Day 169 RF negative | 33 | 40

23. Secondary Outcome: Open-Label LT Period: Number of Participants Achieving ACR 20 Response at Days 169, 729, 1261, and 1821
Description: as for outcome 1
Time Frame: Days 169, 729, 1261, 1821
Population: All participants who entered the LT period and received at least 1 dose of study drug during the LT period were summarized.
Measure: Number; unit: participants
Groups:
- Open-Label SC Abatacept Long Term Period: During the Open-Label LT Period, participants could either continue with or switch to 125 mg weekly SC abatacept injections until the SC formulation became commercially available on a country basis or the Sponsor terminated the study. The Anti-TNF Sub-study terminated due to low recruitment and participants were permitted to roll into the LT Open Label Period.
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1357
participants
  Day 169 (n=1357) | 1087
  Day 729 (n=1187) | 973
  Day 1261 (n=1068) | 904
  Day 1821 (n=421) | 356

24. Secondary Outcome: Open-Label LT Period: Number of Participants Achieving ACR 50 and ACR 70 Responses at Days 169, 729, 1261, 1821
Description: as for outcome 2
Time Frame: Days 169, 729, 1261, 1821
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1362
participants
  Day 169 ACR 50 (n=1362) | 724
  Day 729 ACR 50 (n=1185) | 720
  Day 1261 ACR 50(n=1069) | 672
  Day 1821 ACR 50 (n=423) | 277
  Day 169 ACR 70 (n=1362) | 371
  Day 729 ACR 70 (n=1186) | 443
  Day 1261 ACR 70 (n=1070) | 438
  Day 1821 ACR 70 (n=425) | 191

25. Secondary Outcome: Open-Label LT Period: Mean Change From Baseline in Disease Activity Score in 28 Joints (DAS28) Using C-reactive Protein (CRP) at Days 169, 729, 1261, 1821
Description: The DAS28 index measures disease activity in rheumatoid arthritis and is a composite derived from the number of swollen/tender joints, laboratory tests of inflammation (C-reactive protein measured in mg/L), and participant assessment of global health (by marking a visual analog scale 100 mm line from "very good" to "very bad"). A higher DAS28 score indicates worse control of disease. High disease activity is > 5.1, low disease activity is < 3.2 and remission is < 2.6. A clinically significant response= decrease in DAS28 score of >1.2 from baseline.
Time Frame: Days 169, 729, 1261, 1821
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1353
units on a scale
  Day 169 (n=1353) | -2.65 [-2.71 to -2.58]
  Day 729 (n=1181) | -2.94 [-3.01 to -2.86]
  Day 1261 (n=1063) | -3.09 [-3.17 to -3.00]
  Day 1821 (n=413) | -3.24 [-3.38 to -3.11]

26. Secondary Outcome: Open-Label LT Period: Number of Participants Achieving DAS 28 Remission at Days 169, 729, 1261, 1821
Description: The DAS28 index measures disease activity in rheumatoid arthritis and is a composite derived from the number of swollen/tender joints, laboratory tests of inflammation (C-reactive protein measured in mg/L), and participant assessment of global health (by marking a visual analog scale 100 mm line from "very good" to "very bad"). A higher DAS28 score indicates worse control of disease. High disease activity is > 5.1, low disease activity is < 3.2 and remission is < 2.6.
Time Frame: Days 169, 729, 1261, 1821
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1355
participants
  Day 169 (n=1355) | 334
  Day 729 (n=1183) | 411
  Day 1261 (n=1064) | 425
  Day 1821 (n=413) | 169

27. Secondary Outcome: Open-Label LT Period: Number of Participants Achieving DAS 28 Low Disease Activity (LDA) at Days 169, 729, 1261, 1821
Description: as for outcome 26
Time Frame: Days 169, 729, 1261, 1821
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1355
participants
  Day 169 (n=1355) | 553
  Day 729 (n=1183) | 600
  Day 1261 (n=1064) | 585
  Day 1821 (n=413) | 238

28. Secondary Outcome: Open-Label LT Period: Number of Participants With HAQ-DI Response at Days 169, 729, 1261, 1821
Description: The disability section of the full HAQ includes 20 questions to assess physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do. HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. HAQ-DI overall score ranges from a minimum of 0 to a maximum of 3.0. HAQ response was defined as an improvement (reduction) from baseline (Day 1) of at least 0.3 units in the HAQ score.
Time Frame: Days 169, 729, 1261, 1821
Population: All participants who entered the LT period, received at least 1 dose of study drug during the LT period, and had HAD-QI scores at baseline and at specified days were summarized.
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1364
participants
  Day 169 (n=1364) | 962
  Day 729 (n=1190) | 853
  Day 1261 (n=1068) | 780
  Day 1821 (n=427) | 315

29. Primary Outcome: Anti-TNF Failure Sub-Study Double Blind Period : Number of Participants With Positive Anti-abatacept or Anti-Cytotoxic T Lymphocyte Antigen 4-T Cell (CTLA4-T) Response in Anti-TNF Failure Population
Description: Serum samples from all treated adult participants with active rheumatoid arthritis who were from the Anti-TNF failure population were screened for the presence of drug-specific antibodies using Enzyme Linked Immunoabsorbant Assay (ELISA). The number of participants who had the presence of anti-abatacept antibodies or anti-CTLA-4 antibodies present in their serum are summarized.
Time Frame: Days 85, and 169 and postvisits on Days 28, 56, and 85
Population: All randomized participants in the Anti-TNF Failure Sub-study who received at least 1 dose of study medication. n=Number of participants with at least 1 assessment available.
Measure: Number; unit: participants
Groups:
- Subcutaneous Abatacept: Participants received weekly injections of 125 mg subcutaneous abatacept (with a loading dose of intravenous (IV) abatacept on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV placebo) with the exception that on Day 1, a loading dose of IV abatacept replaced the IV placebo treatment. An Anti-TNF Failure Sub-study was initiated using the same treatment as the Main study in order to assess the immunogenicity and safety in the Anti-TNF Failure population.
- Intravenous Abatacept: Participants received IV abatacept infusions on Days 1, 15, and 29 and every 28 days thereafter. A double-dummy design was used to protect the blind, thus, participants also received subcutaneous injections of placebo (subcutaneous placebo). An Anti-TNF Failure Sub-study was initiated using the same treatment as the Main study in order to assess the immunogenicity and safety in the Anti-TNF Failure population.
Arm/Group | Subcutaneous Abatacept | Intravenous Abatacept
Number analyzed (Participants) | 8 | 10
participants
  Day 85 Anti-abatacept (n=8,10) | 0 | 0
  Day 85 Anti-CTLA4-T (n=8,10) | 0 | 0
  Day 169 Anti-abatacept (n=6,9) | 0 | 0
  Day 169 Anti-CTLA4-T(n=6,9) | 1 | 0
  Overall Treatment Anti-abatacept (n=8,10) | 0 | 0
  Overall on Treatment Anti-CTLA4-T(n=8,10) | 1 | 0
  28 days post Anti-abatacept (n=1,1) | 0 | 0
  28 days post Anti-CTLA4-T (n=1,1) | 0 | 0
  56 days post Anti-abatacept (n=0,1) | 0 | 0
  56 days post Anti-CTLA4-T (n=0,1) | 0 | 0
  85 days post Anti-abatacept (n=0,1) | 0 | 0
  85 days post Anti-CTLA4-T (n=0,1) | 0 | 0

30. Secondary Outcome: Open-Label LT Period: Number of Participants With Death As Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Treatment-related AEs, or AEs Leading to Discontinuation
Description: as for outcome 6
Time Frame: End of ST Period (Day 169) to last dose plus 85 days, up to 5 years (September 2014)
Population: All participants who entered the LT Period and received at least 1 dose of study drug during the LT Period.
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1373
participants
  Death | 41
  SAE | 353
  Treatment-related SAE | 88
  SAEs leading to Discontinuation | 73
  Treatment-related AEs | 632
  AEs leading to Discontinuation | 97

31. Secondary Outcome: Open-Label LT Period: Number of Participants With AEs of Special Interest
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs: all infections, serious infections, and opportunistic infections; autoimmune disorders; malignancies; system injection reactions, and local injection site reactions.
Time Frame: End of ST Period (Day 169) to last dose plus 85 days, up to 5 years (September 2014)
Population: All participants who entered the LT Period and received at least 1 dose of study drug during the LT Period.
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1373
participants
  All Infections | 962
  Serious Infections | 85
  Infections leading to Discontinuation | 25
  Serious Infections leading to Discontinuation | 16
  Malignancies | 56
  Autoimmune Disorders | 67
  Local Injection Site Reactions | 33
  Systemic Injection Reactions | 161

32. Secondary Outcome: Open-Label LT Period: Number of Participants With Clinically Significant Abnormalities in Vital Sign Measurements
Description: Vital sign assessments were performed in the LT period at 12-week intervals and at a yearly visit (at 16-week intervals) and, for participants who withdrew from the study prematurely, 7 days after the last dose of SC abatacept. Vital signs included seated systolic blood pressure, seated diastolic blood pressure, temperature, and heart rate. Abnormalities were determined to be clinically significant by the investigator.
Time Frame: End of ST Period (Day 169) to last dose plus 7 days, up to 5 years (September 2014)
Population: All participants who entered the LT Period and received at least 1 dose of study drug during the LT Period.
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1373
participants | 0

33. Secondary Outcome: Open-Label LT Period: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory assessments were performed in the LT period at 12-week intervals and at a yearly visit and, for participants who withdrew from the study prematurely, 7 days after the last dose of SC abatacept. Abnormalities were determined to be clinically significant by the investigator.
Time Frame: End of ST Period (Day 169) to last dose plus 7 days, up to 5 years (September 2014)
Population: All participants who entered the LT Period and received at least 1 dose of study drug during the LT Period.
Measure: Number; unit: participants
Arm/Group | Open-Label SC Abatacept Long Term Period
Number analyzed (Participants) | 1373
participants | 0

ADVERSE EVENTS:
Time Frame: First dose (Day 1) in ST period to last dose in LT period plus 85 days, up to 5 years (September 2014).
Description: Population includes both Main Study and Anti-TNF Failure Sub-study. Sub-study was terminated early and participants could enter LT Period of Main study.
Groups:
- IV Abatacept: During the Main study Double Blind ST Period, participants received IV abatacept infusions on Days 1, 15, 29, and every 28 days, thereafter for 6 months. A double-dummy design was used to protect the blind, thus, participants also received SC injections of placebo (SC Placebo). An Anti-TNF Failure Sub-study was initiated (recruited separately from Main study) using the same treatment as the Main study in order to assess the immunogenicity and safety in the Anti-TNF Failure population. The Sub-study terminated due to low recruitment and participants were permitted to roll into the LT Open Label Period. During the Open Label LT Period, participants in both the Main Study and the Anti-TNF Failure Sub-study could switch to SC abatacept until the SC formulation became commercially available on a country basis or the Sponsor terminated the study.
- SC Abatacept: During the Main Study Double Blind ST Period, participants received 125 mg weekly SC abatacept injections for 6 months (with an IV abatacept loading dose on Day 1, based on weight). A double-dummy design was used to protect the blind, thus, participants also received IV injections of placebo (IV Placebo) with the exception that on Day 1 a loading dose of IV abatacept replaced the IV Placebo treatment. An Anti-TNF Failure Sub-study was initiated (recruited separately from Main study) using the same treatment as the Main study in order to assess the immunogenicity and safety in the Anti-TNF Failure population. The Sub-study terminated due to low recruitment and participants were permitted to roll into the LT Open Label Period. During the Open Label LT Period, participants in both the Main Study and the Anti-TNF Failure Sub-study could continue SC abatacept until the SC formulation became commercially available on a country basis or the Sponsor terminated the study.
Arm/Group | IV Abatacept | SC Abatacept
Serious Adverse Events (participants affected / at risk) | 206/731 | 199/744
Other Adverse Events (participants affected / at risk) | 544/731 | 567/744
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Abatacept (N=731) | SC Abatacept (N=744)
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Chest pain (General disorders) | 6 | 4
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Hypersplenism (Blood and lymphatic system disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0
Infective tenosynovitis (Infections and infestations) | 2 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Salpingitis (Infections and infestations) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 4
Urosepsis (Infections and infestations) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3
Basilar migraine (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Jaundice hepatocellular (Hepatobiliary disorders) | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Macular fibrosis (Eye disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Peritoneal tuberculosis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Adhesion (General disorders) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 3
Bacteraemia (Infections and infestations) | 0 | 1
Blindness (Eye disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Cellulitis (Infections and infestations) | 1 | 2
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 4
Drug abuse (Psychiatric disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Enterococcus test positive (Investigations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 2
H1N1 influenza (Infections and infestations) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 2
Mastitis (Infections and infestations) | 1 | 0
Median nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Quadriparesis (Nervous system disorders) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1
Embedded device (General disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 2 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Necrotising granulomatous lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 2 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 2
Renal injury (Renal and urinary disorders) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Uterine prolapse (Reproductive system and breast disorders) | 1 | 2
Viral hepatitis carrier (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Asthenia (General disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metatarsus primus varus (Congenital, familial and genetic disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Mucoepidermoid carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia (Infections and infestations) | 12 | 8
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 2
Schizophrenia (Psychiatric disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Venous thrombosis (Vascular disorders) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 3
Calculus bladder (Renal and urinary disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Device failure (General disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 2
Incarcerated hernia (General disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Multi-organ failure (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 16
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Retinal infarction (Eye disorders) | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Aortic aneurysm (Vascular disorders) | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 2
Chronic sinusitis (Infections and infestations) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Encephalopathy (Nervous system disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 1
Meniere's disease (Ear and labyrinth disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pacemaker generated arrhythmia (General disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 3
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Sudden cardiac death (General disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 2 | 2
Vasculitis (Vascular disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 5
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Circulatory collapse (Vascular disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Cystocele (Reproductive system and breast disorders) | 2 | 3
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mammoplasty (Surgical and medical procedures) | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 11
Myocardial ischaemia (Cardiac disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 12 | 14
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Tetanus (Infections and infestations) | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Abatacept (N=731) | SC Abatacept (N=744)
Abdominal pain (Gastrointestinal disorders) | 27 | 39
Depression (Psychiatric disorders) | 40 | 37
Dizziness (Nervous system disorders) | 40 | 37
Abdominal pain upper (Gastrointestinal disorders) | 47 | 43
Hypertension (Vascular disorders) | 85 | 96
Pharyngitis (Infections and infestations) | 80 | 74
Cough (Respiratory, thoracic and mediastinal disorders) | 74 | 72
Gastroenteritis (Infections and infestations) | 48 | 60
Nasopharyngitis (Infections and infestations) | 143 | 149
Anaemia (Blood and lymphatic system disorders) | 26 | 55
Gastritis (Gastrointestinal disorders) | 30 | 40
Headache (Nervous system disorders) | 88 | 86
Influenza (Infections and infestations) | 55 | 51
Sinusitis (Infections and infestations) | 50 | 69
Bronchitis (Infections and infestations) | 120 | 109
Nausea (Gastrointestinal disorders) | 53 | 79
Urinary tract infection (Infections and infestations) | 133 | 150
Diarrhoea (Gastrointestinal disorders) | 89 | 96
Back pain (Musculoskeletal and connective tissue disorders) | 76 | 76
Upper respiratory tract infection (Infections and infestations) | 131 | 130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.